CLINICAL TRIAL: NCT01520038
Title: Feasibility and Phase 1/II Trial of Adjuvant Radiation Therapy for the Treatment of Urothelial Bladder Cancer Using Proton Therapy or IMRT
Brief Title: Adjuvant Proton Therapy or IMRT for the Treatment of Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19811
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Urothelial Carcinoma of the Bladder
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Proton therapy
Radiation: IMRT

SUMMARY:
Invasive urothelial bladder cancer is a common malignancy causing 14,000 deaths annually in the United States. The primary objective of the feasibility/Phase I portion of the study is to establish the feasibility and safety of proton and the safety of IMRT for patients with pure or mixed variant urothelial carcinoma.

DETAILED DESCRIPTION:
Invasive urothelial bladder cancer is a common malignancy causing 14,000 deaths annually in the United States. The primary objective of the feasibility/Phase I portion of the study is to establish the feasibility and safety of proton and the safety of IMRT. Safety will be based on acute toxicity. The primary objective of the phase II study is to generate estimates of the local failure rate for intermediate and high risk patients treated with either proton therapy or IMRT. The study, however, is not explicitly designed to compare outcomes of proton therapy and IMRT. Secondary objectives include further evaluation of acute and late toxicity, quality of life and estimation of overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Pure or mixed variant urothelial carcinoma o Allowable mixed variant subtypes include: squamous differentiation glandular differentiation nested pattern microcystic micropapillary lymphoepthelioma-like plasmacytoid and lymphoma-like sarcomatoid/carcinosarcoma giant cell trophoblastic differentiation clear cell lipid cell undifferentiated Radical cystectomy and pelvic lymph node dissection within the prior 48 weeks Pathologic T3 or higher stage disease, N0-2, M0 (AJCC, 7th Ed., Appendix C) No clinical evidence of residual or recurrent disease based on the following minimum diagnostic work-up within 8 weeks of a patients consent to participate.

  * History and physical examination
  * Chest imaging by x-ray (PA and lateral views) or CT scan (with or without IV contrast);
  * Axial abdominal and pelvic imaging by MRI (preferably with gadolinium)
  * Bone scan
  * Patients with microscopically involved (positive) surgical margins, but no grossly evident residual disease by imaging or physical exam are eligible.

The patient is a candidate for definitive external beam radiotherapy;

* No prior radiotherapy to the region of study;
* No inflammatory bowel disease, active collagen vascular or connective tissue disorders, and no other medical or social contraindications to radiotherapy, as determined by a participating radiation oncologist; Age ³18 years ECOG performance status: 0-2 Concurrent noninvestigational medications will be permitted Informed consent: Patients must have the ability to understand and be willing to sign the study-specific informed consent indicating their understanding of the investigational nature and the risks of this study before any of the protocol related studies are preformed (this does not include routine laboratory testing or imaging studies required to establish study eligibility);

Exclusion Criteria:

* Unstable renal function in the month prior to registration defined as a creatinine rise of 1 mg/dL Prior partial or complete small bowel obstruction either before or after radical cystectomy Prior radiotherapy to the pelvis; o Prior radiation therapy for a different cancer or disease process is allowed, provided there will be no overlap of radiation therapy fields between the participants prior and current course of radiation therapy, radiotherapy was completed more than four weeks from enrolling in this study.

Planned concurrent chemotherapy or other investigational drug to be given with radiation treatments o Prior chemotherapy or investigational drug for bladder cancer or a different cancer is allowed, provided that: The therapy was completed more than two weeks prior to the start of adjuvant pelvic radiation The participant has recovered to Grade 1 toxicity from agents previously administered Subtotal surgical resection with clinically evident residual disease by physical exam or axial imaging.

Prior or concurrent second invasive malignancy other than prostate and non-melanoma skin cancers, unless disease free for a minimum of five years. If a patient had a concurrent prostate cancer, then it must have been resected to negative margins.

Known severe, active co-morbidity, defined as follows:

o Any clinically significant unrelated systemic illness, medical condition, or other factor, which at the discretion of the Principal Investigators, would interfere in the safe and timely completion of study procedures, compromise the patients ability to tolerate the protocol therapy, or is likely to interfere with the study procedures or results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Christodouleas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjuvant Radiation Therapy for the Treatment of Urothelial Bla: Adjuvant Radiation Therapy for the Treatment of Urothelial Bladder Cancer Using Proton therapy or IMRT
Period: Overall Study
Arm/Group | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Applies to Proton only
Time Frame: withion 14 days of estimated date of treatment completion
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla
Number analyzed (Participants) | 2
Participants | 2

2. Primary Outcome: Number of Participants With Adverse Events
Description: Applies to Both Proton and IMRT
Time Frame: within 90 days of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Late toxicty
Time Frame: later than 90 days from start of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Arm/Group | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla (N=2)
Death NOS (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Radiation Therapy for the Treatment of Urothelial Bla (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes